CLINICAL TRIAL: NCT03960983
Title: Evaluation of the Treatment of Halitosis With Photodynamic Therapy in Older Patients With Complete Denture: Protocol for a Randomized, Controlled Trial
Brief Title: Evaluation of the Treatment of Halitosis With Photodynamic Therapy in Older Patients With Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Halitose PT
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2019-05

CONDITIONS: Halitosis
Keywords: Halitosis; photodynamic therapy; elderly; denture
MeSH Terms: conditions — Halitosis | interventions — Therapeutics; Dentures; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderly pacients with complete dentures and Tongue Scraper (Experimental): Treatment with tongue scraper (n = 20). The participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of repeated before these steps
  Interventions: Device: Treatment with tongue scraper; Procedure: Hygiene procedures for the mucosa and dentures
- Elderly pacients with complete dentures and PDT (Active Comparator): Treatment with Photodynamic therapy (n = 20). The participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis and the microbiological analysis will be repeated before these steps
  Interventions: Radiation: Photodynamic Therapy; Procedure: Hygiene procedures for the mucosa and dentures

INTERVENTIONS:
Device: Treatment with tongue scraper — Treatment with tongue scraper. the evaluation of halitosis will be repeated before this step.
  Arms: Elderly pacients with complete dentures and Tongue Scraper
Procedure: Hygiene procedures for the mucosa and dentures — Hygiene procedures for the mucosa and dentures edentulous participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis will be repeated before this step
  Arms: Elderly pacients with complete dentures and Tongue Scraper
Radiation: Photodynamic Therapy — Treatment with Photodynamic therapy. The evaluation of halitosis will be repeated before this step
  Arms: Elderly pacients with complete dentures and PDT
Procedure: Hygiene procedures for the mucosa and dentures — Hygiene procedures for the mucosa and dentures edentulous participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis will be repeated before this step
  Arms: Elderly pacients with complete dentures and PDT

SUMMARY:
Halitosis is the term used to define an unpleasant odor emanating from the mouth. Some lung diseases and diabetes are among the extra-oral causes of this condition. However, no studies have evaluated the causes and treatment of halitosis in the population of older adults with denture. A randomized, controlled trial is proposed. The patients will be divided into 2 groups: G1: older adults who wear complete dentures and will be treater with tongue scraper (n = 20); G2 older adults who wear complete dentures and will be treater with PDT (n = 20). If the halitosis persists, the participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis will be repeated. If the halitosis is resolved, the participants will return after one week for an additional evaluation. This protocol will determine the effectiveness of photodynamic therapy regarding the reduction of halitosis in older adults with complete denture.

DETAILED DESCRIPTION:
Methods:

A single-center, randomized, controlled, single-blind clinical trial was designed in accordance with the criteria recommended for interventional trials in the SPIRIT Statement. The project for the proposed study received approval from the Human Research Ethics Committee of Universidade Nove de Julho.

Selection of individuals - characterization of sample - Two groups will be composed of older adults (60 years or older) in treatment at the dental clinic of Universidade Nove de Julho. After verbal and written explanations of the study, those who agree to participate will sign a statement of informed consent approved by the Human Research Ethics Committee of Universidade Nove de Julho. The study will be conducted in compliance with the precepts stipulated in the Declaration of Helsinki (revised in Fortaleza, Brazil, 2013).

Calculation of sample size - Initially an error err=|(x_1 ) ̅-(x_2 ) ̅ | was established, where the mean values of groups G1 and G2 whose variances are σ_1^2e σ_2^2, respectively. The effect size was calculated by:

effect size=err/√(σ_1^2+σ_2^2 ) If the normal distribution hypothesis is rejected, the sample size should be corrected by approximately 5%.

Observing statistical samples from the reference Mota et al., 2016; to estimate the mean values and sample variance we obtain the following sample sizes for each group:

Sample Size Group Group Sample Size G1 18 G2 18

Inclusion criteria - Men and women aged 60 years or older using complete dentures.

Exclusion criteria - Dentate patients and edentulous with no complete denture hypersensitivity to the photosensitizing agent used in PDT, H2S < 112ppb.

Training and calibration of examiner - An examiner (gold standard) will perform training and calibration exercises to maximize the reproducibility of the measurements. For such, 10 individuals with halitosis will be evaluated using the Oral Chroma® device. These individuals will not participate in the main study. The intraclass correlation coefficient (ICC) will be calculated for the determination of intra-examiner agreement (≥ 0.90) with regard to the halitosis readings.

Randomization - The 40 individuals with complete denture will be randomized in two groups: Group A (20 individuals submitted to treatment with a tongue scraper) and Group B (20 individuals submitted to treatment with PDT). Opaque envelopes will be identified with sequential numbers (1 to 40) and will contain pieces of paper with the information of the corresponding experimental group (A or B). Blocked randomization will be performed in blocks of five patients (eight blocks for both treatments; example of a block: AABAB). The envelopes will be sealed and kept in numerical order in a safe place until the time of the treatments. The randomization and preparation of the envelopes will be performed by a researcher who will not otherwise participate in the study. Randomization will be performed using Microsoft Excel, version 2013.

Characterization of the study - The experimental design will consist of two groups: G1- older adults with halitosis (SH2 ≥ 112 ppb) who wear complete dentures and treatment with a tongue scraper (n = 20); G2- older adults with halitosis (SH2 ≥ 112 ppb) who wear complete dentures and treatment with PDT (n = 20). The evaluation of halitosis will be performed at baseline (1st session), after treatment with a tongue scraper or PDT (1st session) and after one week (2nd session)

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 60 years or older using complete dentures

* • Halitosis positive: ≥ 112 ppbin the gas chromatography test

Exclusion Criteria:

* Dentate patients and edentulous with no complete denture hypersensitivity to the photosensitizing agent used in PDT, H2S < 112ppb

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Halimetry (Gas Chromatography test) | study completion an average of 1 year]
  The portable Oral ChromaTM will be used for the assessment of halitosis. A syringe will be placed in the patient's mouth with the plunger completely inserted and the participant will breathe through the nose with the mouth closed for one minute.The plunger will then be withdrawn to fill the chamber with air. This procedure will be repeated. The gas injection needle will be placed on the syringe and the plunger will be adjusted to 0.5 ml. This air will be injected into the input of the device in a single motion. This procedure will be done before and immediately after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Vale KLD, Horliana ACRT, Romero SDS, Deana AM, Goncalves MLL, Ferrari RAM, Bussadori SK, Fernandes KPS. Evaluation of the treatment of halitosis with photodynamic therapy in older patients with complete denture: Protocol for a randomized, controlled trial. Medicine (Baltimore). 2019 Jul;98(27):e16275. doi: 10.1097/MD.0000000000016275. PMID 31277154